CLINICAL TRIAL: NCT07016607
Title: Feasibility Study to Assess the Safety and Efficacy of the ViTal Peripheral Intravenous Catheter
Brief Title: Vital Peripheral Intravenous Catheter Feasibility
Acronym: ViTAL-PIVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Embrace Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLP-001
Record Dates: First submitted 2025-05-25; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Catheterization, Peripheral Venous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GPIV (Experimental): If the eligibility criteria are fulfilled, up to 4 attempts will be made to achieve successful peripheral intravenous catheterization with the investigational device. All successive attempts will be made at a site different from the one(s) at which access has already failed.
  Interventions: Device: GPIV

INTERVENTIONS:
Device: GPIV — The investigational device is a peripheral intravenous catheter with a passive fully automatic needlestick protection, with a glide-on-contact design of the plastic cannula tip featuring asymmetry, with the negative, convex slope in the plane perpendicular to the longitudinal axis of the tip resulting in bottom part of the cannula being shorter.
  Other Names: ViTal

SUMMARY:
The goal of this clinical trial is to assess the safety and efficacy of ViTal, a peripheral intravenous catheter with a glide-on-contact design of the plastic canula tip, in peripheral intravenous catheterization in individuals requiring intravenous therapy or blood sampling. The main question it aims to answer is:

What is the first attempt success rate of the peripheral intravenous catheterization done using the study device?

Participants will be asked to grade the pain they experienced when attempts were made to insert the study device into their peripheral vein.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥ 18.
2. Requiring blood sample collection (roll-in subjects) or planned for PIVC (analyzable subjects)
3. Signed informed consent.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Requirement for emergent IV placement (patient's condition would be compromised if there is a delay in IV placement).
3. Previous venous grafts or surgery at the target vessel access site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
First attempt success rate | Periprocedural
  Proportion, in percent, of subjects with successful peripheral intravenous catheterization Successful PIVC is defined as withdrawal of non-pulsatile blood or infusion of saline without evidence of extravasation.
  Failed PIVC is defined as extravasation with initial infusion, inability to draw blood, physician or nurse intervention for access or inability to obtain access.

SECONDARY OUTCOMES:
Device- and procedure-related adverse events | Periprocedural
  Incidence of the device- and procedure-related adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Canela, La Romana, Dominican Republic

IPD SHARING:
Plan to Share IPD: No